CLINICAL TRIAL: NCT06787807
Title: Proteomic Analysis of Patients Undergoing Bariatric Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Alvaro Ferraz, Full professor and head of the general surgery service at UFPE, Universidade Federal de Pernambuco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 78992524100005208
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Colon Cancer; Thyroid Cancer; Esophageal Cancer; Pancreatic Cancer; Gastric Cancer; Potmenopausal Breast Cancer; Endometrial Cancer; Liver Cancer; Gallbladder Cancer; Prostate Cancer; Ovarian; Kidney Cancer; Multiple Myeloma; Meningioma; Breast Cancer; Ovarian Cancer
Keywords: obesity; cancer; bariatric surgery; proteomics; biomarkers; mass spectrometry
MeSH Terms: conditions — Obesity; Colonic Neoplasms; Thyroid Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Endometrial Neoplasms; Liver Neoplasms; Gallbladder Neoplasms; Prostatic Neoplasms; Kidney Neoplasms; Multiple Myeloma; Meningioma; Breast Neoplasms; Ovarian Neoplasms; Neoplasms | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- women with insulin resistance (Experimental): An analysis was made of patients with severe steatosis, among patients undergoing bariatric surgery
  Interventions: Procedure: bariatric surgery
- patients with severe steatosis (Experimental): An analysis was made of patients with severe steatosis, among patients undergoing bariatric surgery
  Interventions: Procedure: bariatric surgery
- General patients with insulin resistance (Experimental): An analysis was made of patients, among men and women, with insulin resistance, among patients undergoing bariatric surgery
  Interventions: Procedure: bariatric surgery
- Patients with above average CRP (Experimental): An analysis was carried out of patients with CRP above the average, among patients undergoing bariatric surgery
  Interventions: Procedure: bariatric surgery
- Patients with grade 1 obesity (Experimental): An analysis was made of patients with grade 1 obesity, among patients undergoing bariatric surgery
  Interventions: Procedure: bariatric surgery
- Patients with grade 2 obesity (Experimental): An analysis was made of patients with grade 2 obesity, among patients undergoing bariatric surgery
  Interventions: Procedure: bariatric surgery
- Patients with grade 3 obesity (Experimental): An analysis was made of patients with grade 3 obesity, among patients undergoing bariatric surgery
  Interventions: Procedure: bariatric surgery

INTERVENTIONS:
Procedure: bariatric surgery — sleeve gastrectomy
  Other Names: sleeve gastrectomy

SUMMARY:
The expression of proteins in the blood of obese individuals is different from the expression of proteins in healthy individuals, and is also different in individuals after bariatric surgery. Therefore, this research aims to better understand protein expression in patients indicated for surgical treatment of obesity, evaluating the pre-operative and post-operative status. The objective of this research is to better understand protein expression in patients indicated for surgical treatment of obesity, evaluating the pre-operative and post-surgery status.

DETAILED DESCRIPTION:
The objective of this study is to analyze the Proteomics of obese patients in the preoperative context of bariatric surgery to evaluate which are the up-regulated proteins - potentially related to oncogenic metabolic pathways - and also the down-regulated proteins in the context of obesity - potentially protective in the context of cancer. As well as, evaluate the variation of these proteins, as well as the metabolic pathways with which they are associated, after weight loss promoted by bariatric surgery, in the period of 01 year after this intervention.

The proteomic study will be carried out based on the formation of pools organized based on the patients' pre- and postoperative similarities. Proteomic analyzes will be carried out on a high-performance liquid chromatography system (nanoUPLC) model Acquity Mclass, Waters. Coupled to a Quadrupole Mass Spectrometer-Time of Flight (QToF) Model Sunapt Xs, Waters. Finally, the raw data (raw mass spectra) will be analyzed by the PROGENESIS QI software (Waters) to identify the proteins.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age with a BMI above 35 kg/m² associated with comorbidity or BMI above 40 kg/m² without comorbidities,

Exclusion Criteria:

* Patients with a previous history of cancer;
* Underage patients
* Patients with other diseases predisposing to the development of cancer: cirrhosis, ulcerative colitis, Barrett's esophagus, etc.
* Patients who have previously undergone bariatric surgery;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2025-09-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with reduced initially upregulated oncogenic proteins | 1 year after bariatric surgery
  reduction of proteins potentially involved in oncogenic metabolic pathways, initially upregulated in the context of obesity

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro B Ferraz, Doctor, Principal Investigator — UFPE
Locations (1):
- Hospital das clínicas da UFPE, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
We are still checking pertinent information for sharing